CLINICAL TRIAL: NCT04035850
Title: Vortioxetine for the Treatment of Hoarding Disorder- an Open Label Study
Brief Title: Vortioxetine for the Treatment of Hoarding Disorder
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Noam Soreni (Other)
Responsible Party: Sponsor-Investigator, Noam Soreni, Associate Professor, Principal investigator, St. Joseph's Healthcare Hamilton
Organization: St. Joseph's Healthcare Hamilton (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7206
Record Dates: First submitted 2019-06-17; First posted 2019-07-29 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder | interventions — Vortioxetine

STUDY DESIGN:
Intervention Model Description: Single group, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Vortioxetine PO tablets, 5-20mg Daily
  Interventions: Drug: Vortioxetine Tablets

INTERVENTIONS:
Drug: Vortioxetine Tablets — Strength 5-20 mg
  Other Names: Trintellix

SUMMARY:
The present study is a single-group open-label investigation of the potential efficacy of Vortioxetine for treatment of 30 adult volunteers with Hoarding Disorder (HD) (flexible-dose study, with a target dose range 5-25mg). The proposed study will be the first Vortioxetine study in HD, and conducted at the Anxiety Treatment and Research Clinic (ATRC) Canada's largest academic anxiety clinic, a regional referral center for individuals with HD. The study requires a Letter of No Objection from Health Canada and the study will be approved by Hamilton Integrated Research Ethics Board (HiREB).

DETAILED DESCRIPTION:
Hoarding disorder (HD) is a common and severe new diagnostic category. HD has two core dimensions: difficulty discarding items and the resultant clutter, which may preclude the use of living spaces for their intended. Other HD criteria, distress and impairment, often include unemployment, removal of children, health risks (e.g. infestations, falls, fires, etc.). The estimated prevalence of hoarding is 5.3% in adults and 2% in youth.

Existing treatments of hoarding are only partially effective. Emerging evidence supports the partial efficacy of cognitive behavioral therapy (CBT) in the treatment of HD though, paradoxically, this therapy mostly addresses the excessive attachment to possessions but not the above-identified cognitive deficits. On the other hand, the study of pharmacological treatments for hoarding is in preliminary stages and there currently are no well-validated or official guidelines for the use of psychotropic medications in HD. Given that HD is a highly prevalent and severe condition, there is an urgent need to address this gap in the literature to improve the well-being of patients with the disorder.

Emerging evidence suggests that serotonergic medications may have an important role in the treatment of HD. First, HD is highly comorbid with obsessive-compulsive disorder (OCD) and major depressive disorder (MDD), two disorders that respond well to serotonergic medications. Second, a recent meta analysis of 14 clinical trials suggested that hoarding symptoms had responded to selective serotonin reuptake inhibitor (SSRIs) (i.e., paroxetine and sertraline) and venlafaxine, a serotonin and norepinephrine reuptake inhibitor, with response rates ranging between 37%-76% of participants. Interestingly, this response rate is similar to response rates reported by meta-analyses of the treatment response of OCD to SRIs. However, those findings should be interpreted with caution given the lack of controlled studies and the diagnostic heterogeneity, the latter a result of the diagnostic ambiguity that prevailed prior to the introduction of HD in the fifth version of the Diagnostic and Statistical Manual (DSM-5).

Treatment of hoarding symptoms should ideally target the obsessional aspect of the syndrome (abnormal attachment to possessions), some or all of the identified cognitive deficits and commonly associated comorbidities. Although preoccupation with possessions, an OCD/MDD-like feature of hoarding, can arguably be addressed by the use of Serotonin reuptake inhibitors (SR) medications that are highly effective for the treatment of OCD and MDD , targeting cognitive deficits in hoarding likely requires a different approach and the use of newer generation serotonergic medications.

Vortioxetine is a novel serotonergic antidepressant with a unique pharmacodynamics profile, reported precognitive effects and proven efficacy for the treatment of MDD . Vortioxetine is a 5-HT3, 5-HT7 and 5-HT1D receptor antagonist, 5-HT1B receptor partial agonist, 5-HT1A receptor agonist and serotonin (5-HT) transporter (SERT) inhibitor. There is preliminary evidence that Vortioxetine's unique serotonergic modulation profile may be associated with distinct mechanisms of action at the brain network level. In addition, several studies1 report that Vortioxetine is associated with improved cognitive performance in patients with MDD. These procognitve effects appear to distinguish Vortioxetine from other antidepressant agents. As such, Vortioxetine should be considered a prime candidate for medication trials in HD. To date, however, no studies of vortioxetine in HD have been published.

With this in mind the goal of the present study is to conduct a preliminary, single-group open-label investigation of the potential efficacy of Vortioxetine for treatment of 30 adult volunteers with HD (flexible-dose study, with a target dose range 5-25mg). The proposed study will be the first Vortioxetine study in HD, and conducted at the ATRC Canada's largest academic anxiety clinic, a regional referral center for individuals with HD. The study requires a letter of no objection from Health Canada and the study will be approved by Hamilton Integrated Research Ethics Board (HiREB).

ELIGIBILITY:
Inclusion Criteria:

1. a principal DSM-5 diagnosis of HD
2. SI-R score>=40
3. age between 25-65
4. no other antidepressant use in the 4 weeks that precede the first Vortioxetine dose*
5. ability to provide written informed consent

   * Patients on non-Vortioxetine antidepressant who are willing to participate in the study and meet all other inclusion and exclusion criteria will be offered a 4-week antidepressant wash out period.

Exclusion Criteria:

1. current or past diagnosis of mania/hypo-mania, psychotic disorder or a 1st-degree relative with bipolar disorder or a psychotic disorder
2. past history of behavioural activation or suicidal ideations on antidepressant medication
3. known hypersensitivity to Vortioxetine
4. concomitant use of other antidepressants
5. current participation in CBT for HD or OCD
6. concomitant use of a MAO inhibitor
7. known hepatic insufficiency
8. pregnancy.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Saving-inventory Revised (SI-R) | 12 weeks
  A self report scale.23-item self-report measure comprising three subscales: difficulty discarding, clutter, and excessive acquisition .
  Items on the SI-R are scored between 0 and 4, with higher scores indicating greater hoarding severity. Total score = sum of all items Range = 0-92. A total score of >46 represents clinically significant hoarding
Hoarding cognitions Inventory | 12 weeks
  Saving cognition Inventory A self report scale that measures hoarding related cognitions.24-item self-report measure of hoarding severity.
  Items on the SI-R are scored between 1 and 7, with higher scores representing more severe hoarding symptoms. indicating Total score = sum of all items, Range = 0-168. Mean score in non clinical population - 42, SD-20; mean score in individuals with HD 95.9 , SD=31.0.

SECONDARY OUTCOMES:
Activities of daily life of hoarding (ADL-H) | 12 weeks
  A self report scale to assess hoarding-related functional impairment
  Total score = sum all 15 items after excluding those rated "Not Applicable"; divide the summed score by the number of items given a numerical rating. This will yield an average of all applicable items. Range = 1-5, score greater than 3 suggests marked functional impairment.
Cognitive changes 1 | 12 weeks
  Cambridge cognition tests:
  Cambridge Gambling Task Multitasking Test Spatial span test Stockings of Cambridge Stop Signal Task
Cognitive changes 2 | 12 weeks
  Digit Symbol Substitution Test (DSST)

CONTACTS AND LOCATIONS:
Overall Officials: Noam Soreni, MD, Principal Investigator — McMaster University, St. Joseph's Healthcare, hamilton, Ontario
Locations (1):
- St Joseph Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No